CLINICAL TRIAL: NCT01257672
Title: Oral Ondansetron vs Domperidone for Symptomatic Treatment of Vomiting During Acute Gastroenteritis in Children: Multicentre Randomized Controlled Trial
Brief Title: Symptomatic Treatment of Acute Gastroenteritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other); Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Ronfani Luca, MD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FARM8E53XM; 2010-019787-36 (EudraCT Number)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Gastroenteritis; Vomiting; Acute Gastroenteritis
Keywords: acute gastroenteritis; vomiting; ondansetron; domperidon; symptomatic treatment
MeSH Terms: conditions — Gastroenteritis; Vomiting | interventions — Ondansetron; Domperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ondansetron (Experimental): ondansetron, syrup, 0,15 mg/Kg of body weight, 1 dose
  Interventions: Drug: Ondansetron
- domperidon (Active Comparator): domperidone, syrup, 0,5 mg/Kg of body weight, one dose
  Interventions: Drug: Domperidone
- placebo (Placebo Comparator): placebo, syrup, one dose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ondansetron — ondansetron syrup (0,15 mg/Kg of body weight)
  Other Names: zofran
  Arms: ondansetron
Drug: Domperidone — domperidone syrup (0,5 mg/Kg of body weight)
  Other Names: Motilium
  Arms: domperidon
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
Vomiting in children with acute gastroenteritis is a major factor of failure of oral rehydration therapy. Effective symptomatic treatment of vomiting would lead to an important reduction in the use of Intravenous Fluid Therapy. Available evidence on symptomatic treatment of vomiting shows the efficacy of the most recently registered molecule (ondansetron) but a proper evaluation of antiemetics drugs largely used in clinical practice, such as domperidone, is lacking.

The aim of this multicentre, double-blind randomized controlled trial is to compare the efficacy of ondansetron and domperidone for the symptomatic treatment of vomiting in children with acute gastroenteritis who have failed Oral Rehydration Therapy.

DETAILED DESCRIPTION:
Vomiting in children with acute gastroenteritis (AG) is not only a direct cause of fluid loss but it is also a major factor of failure of oral rehydration therapy (ORT). Physicians who provide care to paediatric patients in the emergency department (ED) usually prescribe intravenous fluid therapy (IVT) for mild or moderate dehydration when vomiting is the major symptom. Thus, effective symptomatic treatment of vomiting would lead to an important reduction in the use of IVT and, consequently, of the duration of hospital stay and of frequency of hospital admission. Available evidence on symptomatic treatment of vomiting shows the efficacy of the most recently registered molecule (ondansetron) but a proper evaluation of antiemetics drugs largely used in clinical practice, such as domperidone, is lacking.

The aim of this multicentre, double-blind randomized controlled trial conducted in paediatric Emergency Departments is to compare the efficacy of ondansetron and domperidone for the symptomatic treatment of vomiting in children with AG who have failed Oral Rehydration Therapy.

The trial results would provide evidence on the efficacy of domperidone, which is largely used in clinical practice despite the lack of proper evaluation and a controversial safety profile, as compared to ondansetron, which is not yet authorized in Italy despite evidence supporting its efficacy in treating vomiting. The trial results would contribute to a reduction in the use of IVT and, consequently, in hospital admissions in children with AG. The design of this RCT, which closely reflect current clinical practice in EDs, will allow immediate transferability of results

ELIGIBILITY:
Inclusion Criteria:

1. age from 1 to 6 years;
2. presumptive clinical diagnosis of acute gastroenteritis in patients with vomiting, with or without diarrhoea;
3. more than three episodes of non-bilious, non-bloody vomiting within the previous 24 hours;

Exclusion Criteria:

1. treatment with antiemetics or antidiarrhoic drugs in the 6 hours prior to access to ED;
2. underlying chronic diseases (eg, malignancy, gastroesophageal reflux, migraine, renal failure, hypoalbuminemia, liver disease);
3. severe dehydration: weight loss>10% or standardized clinical dehydration score >=18 for children aged 12-24 months and >=16 for older children;
4. known hypersensitivity to ondansetron or domperidone;
5. previous enrolment in the study.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 356 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients needing nasogastric or intravenous rehydration after symptomatic oral treatment failure, defined as vomiting or fluid refusal after the second attempt of ORT. | 6 hours

SECONDARY OUTCOMES:
Percentage of subjects needing hospital admission for the same illness; | 48 hours
Percentage of subjects needing observation stay for more than 6 hours for the same illness | 48 hours
Total emesis duration in the 3 allocation groups; | 48 hours
Number of episodes of vomiting in the 3 treatment groups during the follow-up period | 48 hours
Percentage of subjects presenting adverse events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Federico Marchetti, MD, Study Chair — IRCCS Burlo Garofolo; Maurizio Bonati, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (15):
- Italy (15):
  - Dipartimento di Pediatria, Ospedale Castelli, Verbania, Novara
  - Dipartimento di Emergenza Pediatrica, Ospedale Giuseppe Moscati, Avellino
  - Dipartimento di Emergenza Pediatrica, P.O. Spedali Civili, Brescia
  - Divisione di Emergenza Pediatrica, Ospedale Pediatrico A. Meyer, Florence
  - Unità Operativa di Pediatria, Ospedale GB Morgagni, Forlì
  - Divisione di Emergenza Pediatrica, Istituto G. Gaslini, Genova
  - Dipartimento di Pediatrica, Ospedale di Macerata, Macerata
  - Dipartimento di Pediatria, Azienda Policlinico di Modena, Modena
  - Dipartimento di Emergenza Pediatrica, Azienda Ospedaliera - Università di Padova, Padua
  - Dipartimento di Pediatrica, Azienda Ospedaliera- Università di Parma, Parma
  - Dipartimento di Emergenza Pediatrica, Ospedale Pediatrico IRCCS Bambino Gesú, Roma
  - Dipartimento di Emergenza Pediatrica, Ospedale Infantile Regina Margherita, Torino
  - Dipartimento di Pediatria, Ospedale di Treviso, Treviso
  - Dipartimento di Emergenza Pediatrica, Istituto per la l'Infanzia, IRCCS Burlo Garofolo, Trieste
  - Unità di Terapia Intensiva Pediatrica, Ospedale Civile Maggiore, Verona

REFERENCES:
- [Background] Marchetti F, Maestro A, Rovere F, Zanon D, Arrighini A, Bertolani P, Biban P, Da Dalt L, Di Pietro P, Renna S, Guala A, Mannelli F, Pazzaglia A, Messi G, Perri F, Reale A, Urbino AF, Valletta E, Vitale A, Zangardi T, Tondelli MT, Clavenna A, Bonati M, Ronfani L. Oral ondansetron versus domperidone for symptomatic treatment of vomiting during acute gastroenteritis in children: multicentre randomized controlled trial. BMC Pediatr. 2011 Feb 10;11:15. doi: 10.1186/1471-2431-11-15. PMID 21310051